CLINICAL TRIAL: NCT05641181
Title: Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single-dose CRB4101 Tablets in Healthy Adult Subjects
Brief Title: A Trial of CRB4101 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Resources Biopharmaceutical Co., Ltd (Industry)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZhao
Record Dates: First submitted 2022-11-15; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Intervention Model Description: 100mg, 200 mg, 400 mg, 800 mg, 1200 mg, 1600 mg
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- CRB4101 100mg dose group (Experimental): Participants will receive a single oral dose of 100mg of CRB4101
  Interventions: Drug: CRB4101
- CRB4101 200mg dose group (Experimental): Participants will receive a single oral dose of 200mg of CRB4101
  Interventions: Drug: CRB4101
- CRB4101 400mg dose group (Experimental): Participants will receive a single oral dose of400mg of CRB4101
  Interventions: Drug: CRB4101
- CRB4101 800mg dose group (Experimental): Participants will receive a single oral dose of 800mg of CRB4101
  Interventions: Drug: CRB4101
- CRB4101 1200mg dose group (Experimental): Participants will receive a single oral dose of 1200mg of CRB4101
  Interventions: Drug: CRB4101
- CRB4101 1600mg dose group (Experimental): Participants will receive a single oral dose of 1600mg of CRB4101
  Interventions: Drug: CRB4101
- placebo group (Placebo Comparator): Subjects will receive a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CRB4101 — After the participants who signed the informed consent have been screened by the inclusion criteria, those who meet the inclusion criteria and those who do not meet the exclusion criteria will receive the following 6 dose groups in order from low to high:
  100mg, 200 mg, 400 mg, 800 mg, 1200 mg, 1600 mg In each dose group, 8 participants will be enrolled to receive the drug, including 6 receiving CRB4101 tablets and 2 receiving placebo.
  Other Names: Drug intervention
  Arms: CRB4101 100mg dose group; CRB4101 1200mg dose group; CRB4101 1600mg dose group; CRB4101 200mg dose group; CRB4101 400mg dose group; CRB4101 800mg dose group
Drug: Placebo — After the participants who signed the informed consent have been screened by the inclusion criteria, those who meet the inclusion criteria and those who do not meet the exclusion criteria will receive the following 6 dose groups in order from low to high:
  100mg, 200 mg, 400 mg, 800 mg, 1200 mg, 1600 mg In each dose group, 8 participants will be enrolled to receive the drug, including 6 receiving CRB4101 tablets and 2 receiving placebo.
  Other Names: Placebo intervention
  Arms: placebo group

SUMMARY:
The goal of this clinical trial is toevaluate the safety and tolerability of a single dose of CRB4101 tablets in healthy adults . The main questions it aims to answer are:

* [question 1]The pharmacokinetics (PK) and pharmacodynamic dynamics (PD) characteristics of CRB4101 tablets were evaluated in healthy adults after a single administration.
* [question 2]Exploratory analysis of the relationship between serum concentrations of CRB4101 (and its major metabolites, if necessary) and QTc interphase.
* [question 3]Exploratory analysis of the metabolic and excretory characteristics of CRB4101 after a single administration (if necessary)
* [question 4]Exploratory analysis of pharmacokinetic characteristics of major metabolites of CRB4101 (if necessary)
* [question 5]The influence of pharmacogenomics on pharmacokinetic characteristics (if necessary).

After the participants who signed the informed consent have been screened by the inclusion criteria, those who meet the inclusion criteria and those who do not meet the exclusion criteria will receive the following 6 dose groups in order from low to high:

100mg, 200 mg, 400 mg, 800 mg, 1200 mg, 1600 mg

DETAILED DESCRIPTION:
The subjects who signed the informed consent form were screened by the inclusion and exclusion criteria. The subjects who met the inclusion criteria and did not meet the exclusion criteria were treated with 100 mg, 200mg, 400mg, 800 mg, 1200 mg and 1600 mg in order from low to high. In each dose group, 8 subjects will be enrolled to receive CRB4101 tablets (6 subjects) and placebo (2 subjects). In order to ensure the safety of the subjects, the sentinel method was used to enroll the subjects. Two subjects were enrolled in each dose group (1 patient received CRB4101 and 1 patient received placebo), and the safety of the drugs was evaluated at least 24 hours after administration. The remaining 6 subjects (5 to receive CRB4101 tablets and 1 to receive placebo) could be enrolled if the investigator assessed that the subjects had tolerable safety. Therefore, a total of 48 subjects were planned to be recruited for single-dose safety, tolerability, PK, and PD studies. Subjects were admitted to the clinical trial facility 1 day before administration (D-1), fasted for at least 10 h before administration, and received a single oral dose of CRB4101 tablets or placebo on the day of administration (D1). Subjects will be hospitalized for laboratory tests, vital signs, adverse events, safety and tolerability evaluation, and PK and PD samples of CRB4101 tablets will be collected. Subjects will leave the clinical trial facility after completing the safety assessment on the 4th day after administration (D4), return to the clinical trial facility 10 days after departure (D14±1), and leave the clinical trial facility after completing the last safety check (safety follow-up).

The dose was increased from low to high, and each subject could only receive one dose. "When safety data are available for all patients in a dose arm after day 14, the investigator and the sponsor will jointly assess safety, tolerability, and available PK/PD results at that dose level to determine whether to proceed to the next dose arm." If the criteria for dose escalation were met, escalation to the next dose was performed. If the criteria for discontinuation of dose escalation were met, exploration could continue at the reduced dose level after joint review and confirmation by the investigator and sponsor. If after the maximum climbing dose (1600 mg) was reached, the review of human safety data did not meet the stopping criteria, and the investigator and the sponsor jointly decided that further climbing was necessary, the Ethics committee needed to apply for an increase again. If criteria for dose escalation were observed to be met in a given group, the plan would be discontinued. At this point, the investigator and the sponsor could discuss together whether to continue the study with a dose reduction based on available safety, tolerability, PK, and PD data. Option to continue the study at 1000 mg).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants aged between 18 and 50 years (including 18 and 50 years) (the ratio of male/female participants to all is required to be no less than 1/3 in the groups with the dose of 200mg, 400mg and 800mg);
2. Male weight in the range of 50 kg(inclusive) to 90kg, female weight in the range of 45 kg(inclusive) to 90 kg, body mass index (BMI= weight/height square (kg/㎡)) :19.0≤BMI < 28.0;
3. participant who is able to communicate well with the investigator and is willing and able to comply with all planned visits, laboratory examinations, and other study procedures.
4. Have fully understood this study, voluntarily participated in the experiment, and have signed written informed consent form.

Exclusion Criteria:

1. Pregnant, lactating women, or female participants of childbearing potential who have not used contraception for at least 30 days before drug administration; Male participants who are unwilling to use contraception (or could not guarantee not to donate sperm) and female participants of childbearing potential who are unwilling to use contraception during enrollment in the trial and for 90 days after dosing;
2. Suspected or definitely confirmed (inquiry) allergy to the study drug or any component in the study drug, or allergic constitution;
3. participants with diseases or previous diseases (including but not limited to cardiac/cardio-cerebrovascular, respiratory, endocrine, metabolic, renal, hepatic, gastrointestinal, dermatological, malignant, hematological, immune, infectious, neurological or psychiatric diseases), surgical history or any other conditions judged by the investigator to affect the absorption, distribution, metabolism and excretion of drugs or to reduce compliance ;
4. Have a personal or family history of bleeding diseases or coagulopathy, or have long-term or unexplained abnormal bleeding, such as frequent epistaxis (nosebleeds), gum bleeding, or have a high risk of bleeding such as hemorrhoids, gastrointestinal ulcers, or often have unexplained bruises/ecchymosis; participants with definite history of hemoptysis, hematemesis, melena or hematuria; Or women who are expected to be menstruating at the time of administration;
5. History of cerebral hemorrhage (including congenital cerebral vascular malformations such as cerebral arteriovenous malformations or cavernous hemangiomas), stroke, and cerebrovascular accident (CVA)
6. Have had risk factors for torsade de pointes, or have had a first-degree relative (i.e., biological parent, sibling, or child) family history of short QT syndrome, long QT syndrome, unexplained sudden death, drowning, or sudden infant death in young adulthood (less than or equal to 40 years of age);
7. Abnormal and clinically significant hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia or hypocalcemia as judged by the investigator;
8. participants received anticoagulant or antiplatelet therapy within 1 month before screening; Or with adverse reactions of anticoagulant or antiplatelet drugs;
9. participants with severe head trauma or major head surgery within 2 years before screening;
10. Underwent major surgery within 3 months before screening or any surgery within 1 month before screening or plan to undergo surgery within 2 weeks after the end of the study;
11. Individuals who has donated blood within 1 month prior to screening, or donated ≥400 mL of blood within 3 months prior to screening, or received blood or blood component transfusion within 8 weeks prior to screening and before dosing;
12. Taking any prescription drugs, over-the-counter drugs or herbal medicines within 2 weeks before taking the study drug, or within 5 half-lives of the drug at the time of screening;
13. Regular alcohol use in the 3 months before screening (14 units per week: 1 unit = 285 mL of beer; Or liquor 25 mL; Or wine 125 mL), or with abnormal results of alcohol breath test before enrollment;
14. Smoking (≥5 cigarettes per day) or using smoking cessation products or nicotine-containing products within 2 weeks before taking the study drug; Or unable to stop using any tobacco-based products after enrollment throughout the trial;
15. participants with glucose intolerance or rare genetic diseases - galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption;
16. Consuming grapefruit/grapefruit/grapefruit, coffee, tea, and other foods or beverages containing caffeine or alcohol within 7 days before taking the study drug; Or strenuous exercise; Or have special requirements for diet, can not abide by the uniform diet;
17. There are clinically significant abnormalities in vital signs, physical examination, 12-lead electrocardiogram, chest X-ray, abdominal ultrasound, and laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function, fecal occult blood).
18. The results of APTT, PT or INR at screening/baseline are beyond the normal range and confirmed by repeated tests;
19. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or gamma-glutamyltransferase (GGT) above the upper limit of normal (ULN), or total bilirubin >ULN, or lipase or amylase >ULN at screening/baseline visit;
20. Serum creatinine >ULN at screening/baseline visit;
21. During the screening period, infectious diseases are screened for any positive of hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody (anti-HCV), human immunodeficiency virus (HIV) antibody and syphilis antibody.
22. Stool occult blood test is positive before randomization;
23. History of drug abuse or positive urine drug screening at screening/baseline visit;
24. participants who have participated in a clinical trial within 3 months before screening;
25. Those who are not suitable for venous blood collection;
26. Any other circumstances in which the participant are deemed by the investigator to be ineligible for the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-04-05 (Estimated); Study Completion 2023-06-21 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study (approximately 20 days)
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-Tmax | Up to 3 days
  Time to reach Cmax for CRB4101 and its metabolites
Pharmacokinetics-Cmax | Up to 3 days
  Peak concentrations of CRB4101 and its metabolites were observed
Pharmacokinetics-AUC0- 24h | Up to 3 days
  Area under the concentration-time curve from time 0 to 24h after CRB4101 administration
Pharmacokinetics-AUC0-t | Up to 3 days
  Area under the concentration-time curve from time 0 to t after CRB4101 administration
Pharmacokinetics-AUC0-∞ | Up to 4 days
  Area under the concentration-time curve from time 0 to ∞ after CRB4101 administration
Pharmacokinetics-Vd/F | Up to 3 days
  Area under the concentration-time curve from time 0 to t after CRB4101 administration
Pharmacokinetics-CL/F | Up to 3 days
  Plasma clearance of CRB4101 and its metabolites
Pharmacokinetics-t1/2 | Up to 3 days
  Plasma elimination half-life of CRB4101 and its metabolites
Pharmacokinetics-Kel | Up to 3 days
  CRB4101 and its metabolite terminal elimination rate constants
Pharmacokinetics-MRT | Up to 3 days
  Mean retention time of CRB4101 and its metabolites
Pharmacokinetics-Ae | Up to 3 days
  Cumulative urinary excretion of CRB4101 and its metabolites
Pharmacokinetics-CLr | Up to 3 days
  Renal clearance of CRB4101 and its metabolites
Pharmacokinetics-Fe | Up to 3 days
  Cumulative excretion rates of CRB4101 and its metabolites
Pharmacodynamics-APTT | Up to 20 days
  APTT
Pharmacodynamics-PT | Up to 20 days
  PT
Pharmacodynamics-INR | Up to 20 days
  INR
Pharmacodynamics-FXI：C | Up to 20 days
  FXI：C
Pharmacodynamics-Coagulation factor XIa activity. | Up to 20 days
  Coagulation factor XIa activity
Pharmacodynamics-QTc | Up to 3 days
  QTc

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No